CLINICAL TRIAL: NCT06928298
Title: Cognitive Screening Made Easy for PCPs - Administrative Supplement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Robin C. Hilsabeck, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AG069780-04S
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cognitive Impairment; Cognitive Decline; Dementia, Mild
Keywords: older adults; mild cognitive impairment; mild dementia; cognitive screening; primary care; dementia screening
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Risk assessment and cognitive screening app that includes questions answered by the participant and completion of a working memory task and two speech tasks
  Interventions: Behavioral: RACS app

INTERVENTIONS:
Behavioral: RACS app — risk assessment questions, symbol matching task, voice tasks

SUMMARY:
This project will facilitate early detection of cognitive decline in older adults through development and implementation of an automated risk assessment and cognitive screening tool for use in primary care. By providing an automated tool developed specifically to address the needs of PCPs, it will be easier to screen for cognitive impairment, increasing the number of older adults who are screened and thus identified and treated.

DETAILED DESCRIPTION:
In the United States and around the world, people are living longer lives. As the population ages, so does the number of older adults who may experience declines in memory, attention, reasoning, or other thinking skills. Some of these changes in cognition can be treated and reversed if caught early. Others can be slowed down and hopefully one day prevented. Unfortunately, people with cognitive decline or very mild dementia often are not recognized until late in the disease course when treatments are less effective. As the first health care professional most people reach out to about medical concerns, primary care providers play a critical role in detecting cognitive decline early. While many primary care providers conduct cognitive screening at Medicare Annual Wellness Visits and when patients voice concerns, 9 out of 10 would like more information about who to screen, which assessment tool to use, and what to say if screening is positive. Deciding who to screen with a brief cognitive assessment tool is a key part of the process because not everyone needs to be screened, and primary care providers already face time pressures to address the obvious and immediate concerns of their patients. The long-term goal of this project is to develop a risk assessment and cognitive screening tool that requires minimal time and effort from primary care providers or their staff and is sensitive to cognitive decline in older adults from diverse educational and racial/ethnic backgrounds. The tool will be integrated into electronic health record systems to make it easy for primary care providers and patients to see results. The specific aims for the administrative supplement of the R33 phase of this project are to further test the effectiveness of the newly developed risk assessment and cognitive screening application in 100 Spanish speaking older adults receiving care in primary care clinics, to find out from primary care providers using the tool how much they liked it and if it was useful and easy to use, and to integrate findings into multiple electronic health record systems. Findings from this project will fill a gap in the existing toolkit of primary care providers and will make screening for cognitive decline quick, easy, effective and accessible in more than one language.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Aged 60 years and older;
* Ethnic/racial background consistent with NIH policy
* Male or female
* Fluent in Spanish.

Exclusion Criteria:

* Confounding conditions that could impact ability to participate in the study (e.g., cognitive impairment sufficient to impact ability to follow instructions on the iPad, motor impairment that would prohibit independent use of RACS, poor visual acuity)
* Prior diagnosis of dementia
* Non-Spanish speaking.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance Score | baseline, 6 month, and 12 month visits
  Combination of symbol matching and voice tasks, which generates a cognitive performance score ranging from 0 to 1 (high scores mean higher likelihood of cognitive impairment)

SECONDARY OUTCOMES:
Usability | baseline, 6 month, and 12 month visits
  Questions about usability completed by clinic staff and PCPs. The scale is a modified version of the Usefulness, Satisfaction, and Ease of Use (USE) questionnaire. Scores range from 8 to 56, with higher scores indicative of greater usability.

CONTACTS AND LOCATIONS:
Overall Officials: Robin C Hilsabeck, PhD, Principal Investigator — University of Texas Health Sciences Center at San Antonio
Locations (3):
- United States (3):
  - Family Wellness Clinic, Austin, Texas
  - University of Texas Health Austin Primary Care Clinic, Austin, Texas
  - UT Health San Antonio's Geriatrics and Supportive Care Clinic, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include demographic and clinical data, scores on neuropsychological tests, speech samples, and machine learning algorithms.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Release of the final data and RACS app will be made available by the online publication date
Access Criteria: The investigators will publish all of the code and scripts for statistical analysis and machine learning development on a publically available GitHub repository.